CLINICAL TRIAL: NCT04979013
Title: BRP1802 Changes in Biomarkers of Potential Harm Over Two Weeks of Smoking Abstinence
Brief Title: BRP1802 Smoking Abstinence Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BRP1802
Record Dates: First submitted 2021-05-11; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Smoking; Smoking Cessation; Tobacco Use
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smoking Abstinence (Experimental): 14-day Smoking Abstinence
  Interventions: Other: Smoking Abstinence

INTERVENTIONS:
Other: Smoking Abstinence — Smokers will be switched to smoking abstinence for 14 days

SUMMARY:
A single-center study designed to evaluate changes in short-term biomarkers of potential harm (BoPH) in healthy adult cigarette smokers of two age groups (Group A: 24-34 years; Group B: 35-60 years) during 14 days of smoking abstinence.

DETAILED DESCRIPTION:
The overall goal of the smoking abstinence study is to discover and assess biomarkers that respond rapidly to smoking abstinence and explore whether the smokers' age influences the responsiveness of biomarkers to changes in smoking status. The study is a single-center, parallel cohort, in which generally healthy adult male and female smokers participated. Smokers of 10-30 cigarettes per day for at least 5 years prior to screening were recruited. Plasma and urine (24h and spot urine) samples and other biological specimens will be collected at the baseline and at specified timepoints during the course of the study. The study will include two primary study cohorts, smokers ages 24-34 years and 35-60 years, to determine whether age could be a confounder in the qualification of biomarkers. Starting on Day -2, eligible smokers will be confined at the clinical site for 17 days. Biological samples will be collected on Days -2 and -1 for baseline study endpoints. On Day 1, smokers will be switched to smoking abstinence for 14 days. Samples will be collected for endpoint analysis throughout the 14-day abstinence period.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy male or female adults, 24 to 60 years of age, inclusive, at the time of consent.
3. Able to safely perform the required study procedures, as determined by the Investigator.
4. Exhaled carbon monoxide (ECO) level is ≥ 10 ppm and ≤ 100 ppm at Screening and Day -2.
5. Positive urine cotinine test at Screening and Day -2.
6. Smokes only combustible, filtered, non-menthol or menthol cigarettes, 83 mm to 100 mm in length.
7. Agrees to smoke same Usual Brand (UB) cigarette on Days -2 and -1. UB cigarette is defined as the cigarette brand style currently smoked most frequently by the subject.
8. Smokes 10-20 combustible filtered cigarettes per day and inhales the smoke, and has smoked for at least 5 years prior to Screening. Brief periods of abstinence due to illness, quit attempt (30 days prior to Enrollment), or clinical study participation (30 days prior to Enrollment) will be allowed at the discretion of the Investigator. Occasional usage of other tobacco or nicotine containing products may be allowed at the discretion of the Sponsor.
9. Willing to abstain from smoking during the study's abstinence period.
10. Females must be willing to use a form of contraception acceptable to the Investigator from the time of signing informed consent until Study Discharge.

    Forms of contraception are:
    * Sexually inactive (abstinent as a lifestyle) for 28 days prior to Day -2. A female subject who claims to be sexually inactive but becomes sexually active during the course of the study, must agree to use a physical barrier method (e.g., condom, diaphragm) with spermicide from the time of the start of sexual activity and throughout the study.
    * Using birth control methods:

      * hormonal oral contraceptives, vaginal ring, transdermal patch, or hormone or non-hormone releasing intrauterine device for at least 3 months prior to Day -2 and throughout the study.
      * depot/implantable hormone (e.g., Depo-provera®, Implanon) for at least 3 months prior to Day -2 and throughout the study.
      * surgical sterilization of the partner (vasectomy for 4 months minimum) prior to Day -2.
      * physical barrier method (e.g., condom, diaphragm) with spermicide for at least 14 days prior to Day -2 and throughout the study.
    * Have undergone one of the following sterilization procedures at least 6 months prior to Day -2:

      * hysteroscopic sterilization
      * bilateral tubal ligation or bilateral salpingectomy
      * hysterectomy
      * bilateral oophorectomy
11. Agrees to in-clinic confinement of 17 days and 16 nights.
12. Agrees to have samples collected and stored for future use.

Exclusion Criteria:

1. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the Investigator, makes the study participant unsuitable to participate in this clinical study.
2. History, presence of, or clinical laboratory test results indicating diabetes.
3. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes.
4. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As needed treatment, such as inhalers, may be included at the Investigator's discretion pending approval from the Medical Monitor.
5. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
6. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
7. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to the signing of informed consent.
8. Use of medication that impacts lung function biomarkers or other biomarkers within 2 weeks of study enrollment (i.e., Day -2), including acetylsalicylic acid (Aspirin) or ibuprofen and antibiotics. After enrollment, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the Investigator or designee.
9. Participation in another clinical trial within (≤) 30 days prior to the signing of informed consent. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing informed consent in the current study.
10. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
11. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
12. A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at Screening and Day -2.
13. Drinks more than 21 servings of alcoholic beverages per week or has a positive alcohol result at Screening and Day -2.
14. Hemoglobin level is < 12.5 g/dL for females or < 13.0 g/dL for males at the Screening Visit;
15. History or presence of bleeding or clotting disorders;
16. Any use of anticoagulants;
17. Whole blood donation within eight weeks (≤ 56 days) prior to the signing of informed consent;
18. Plasma donation within (≤) seven days prior to the signing of informed consent;
19. Weight of ≤ 110 kg;
20. Employed by a tobacco or nicotine company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
21. Determined by the Investigator to be inappropriate for this study.

Ages: 24 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Urinary Arachidonic Acid (AA) Metabolites 2,3-dinor-thromboxane B2 (TxM) and leukotriene E4 (LTE4) | 14 days
  Change in Urinary Arachidonic Acid (AA) Metabolites TxM and LTE4

SECONDARY OUTCOMES:
Urinary AA metabolites TxM and LTE4 | 7 days
  Change in Urinary AA metabolites TxM and LTE4
Additional AA metabolites | 14 days
  Change in additional AA metabolites:
  Tetranor-prostaglandin (t-PGDM); Tetranor-prostaglandin E metabolite (t-PGEM); 2,3-dinor-8-iso prostaglandin F2alpha (2,3-d-8-iso-PGF2α); 8-iso prostaglandin F 2alpha (8-iso-PGF2α); Prostaglandin F 2alpha (PGF2α); 11-dehydrothromboxane B2 (11-dh-TXB2); 20-carboxy-leukotriene B4 (20-COOH-LTB4); 20-hydroxy-leukotriene B4 (20-OH-LTB4)
Biomarkers of Exposure in Urine: Nicotine equivalents and CEMA | 14 days
  Change in biomarkers of exposure in Urine:
  Nicotine equivalents (molar sum of nicotine + 5 metabolites); 2-cyanoethylmercapturic acid (CEMA)
Biomarkers of Exposure in Urine: TSNAs | 14 days
  Change in biomarkers of exposure in Urine:
  Tobacco Specific Nitrosamine(s) (TSNAs)
Biomarkers of Exposure in Blood: Carboxyhemoglobin | 14 days
  Change in biomarkers of exposure in Blood:
  Whole blood carboxyhemoglobin
Biomarkers of Exposure in Blood: nicotine and cotinine | 14 days
  Change in biomarkers of exposure in Blood:
  Plasma nicotine; Plasma cotinine
Biomarkers of Potential Harm: FeNO | 14 days
  Change in biomarkers of potential harm:
  Fractional expired Nitric Oxide (FeNO)
Biomarkers of Potential Harm: ABG | 14 days
  Change in biomarkers of potential harm:
  Arterial Blood Gas (ABG)
Nasal Mucociliary Clearance (NMC) Saccharin Transit Time (STT) | 14 days
  Change in Nasal Mucociliary Clearance (NMC) Saccharin Transit Time (STT)
T- and B-lymphocytes and Natural Killer (NK) cell profiles | 14 days
  Change in T- and B-lymphocytes and Natural Killer (NK) cell profiles
Changes in Platelet Aggregation | 14 days
  Evaluation of platelet aggregation using Adenosine Diphosphate (ADP) as an agonist from baseline to Day 14. Platelet aggregation testing measures the ability of various agonists to platelets to induce ex vivo activation and platelet-to-platelet activation.

CONTACTS AND LOCATIONS:
Overall Officials: Bobbette Jones, DrPH, Study Director — RAIS
Locations (1):
- Celerion Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No